CLINICAL TRIAL: NCT01174433
Title: Safety Study to Assess the FEasibility of Use of the TRYTON Bifurcation Coronary Stent System (SAFE-TRY)
Acronym: SAFE-TRY
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Mirano's Hospital, Mirano, Italy (Unknown); San Giacomo Apostolo Hospital, Castelfranco Veneto, Italy (Unknown); Conegliano Veneto's Hospital, Conegliano Veneto, Italy (Unknown)
Responsible Party: Principal Investigator, Giuseppe Tarantini, MD, PhD, University of Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2040P
Record Dates: First submitted 2010-07-28; First posted 2010-08-03 (Estimated); Last update posted 2012-07-04 (Estimated); Status verified 2012-07

CONDITIONS: Coronary Artery Disease; Angioplasty, Transluminal, Percutaneous Coronary
Keywords: Bifurcation coronary artery disease; Percutaneous coronary intervention; Tryton Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tryton bifurcation stent system (Experimental)
  Interventions: Device: Tryton

INTERVENTIONS:
Device: Tryton — Percutaneous coronary intervention of a bifurcation lesion, with a Tryton bifurcation coronary stent for the side branch and a drug-eluting coronary stent for the main branch
  Other Names: Tryton bifurcation stent system

SUMMARY:
To assess the safety and feasibility of the use of the Tryton bifurcation coronary stent system for the treatment of single de novo bifurcation lesions in native coronary arteries.

DETAILED DESCRIPTION:
Currently available stents were designed for straight lesions, optimised to provide scaffolding (coverage and radial strength) and ease of deliverability. In straight lesions, these stents have been shown to provide superb acute and long-term results. One lesion subset that continues to challenge the interventionalist is bifurcations lesions. A number of different strategies have been employed with standard stents to address bifurcation lesions each of which have significant limitations. Large contemporary registries characterising current stent usage in bifurcating lesions have demonstrated decreased procedural success with increased rates in restenosis and thrombosis (acute, subacute and delayed). The limitations of currently available stents have led groups to develop stents designed specifically to treat bifurcation lesions. The Tryton Side-Branch Stent Stent TM (Tryton Medical, Inc., Newton, MA, USA) is a balloon expandable cobalt chromium stent, designed specifically to treat bifurcation lesions.

The primary objective of this study is to evaluate the safety and feasibility of the use of the Tryton bifurcation coronary stent system for the treatment of single de novo bifurcation lesions in native coronary arteries with reference vessel diameters (RVD) for the proximal main vessel of 2.5 - 5.0 mm, distal main branch of 2.5 - 5.0 mm, and side branch RVD 2.5 - 3.5 mm.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

* Candidate for percutaneous coronary intervention & emergent coronary artery bypass graft surgery
* Clinical evidence of ischemic heart disease or a positive functional study
* Female patients of childbearing potential has negative pregnancy test within 7 days before trial procedure
* Patient or patient's legal representative provided written informed consent
* Patient agrees to comply with follow-up evaluations

Angiographic Inclusion Criteria

* Target lesion in a single de novo true bifurcation lesion (Medina classification Type 1.1.1; 1.0.1; 0.1.1; 0.0.1) involving a native coronary artery with reference vessel diameter for the proximal main of 2.5 - 5.0 mm, distal main of 2.5 - 5.0 mm, & side branch RVD of 2.5 - 3.5 mm
* Target lesion in main vessel has stenosis of > 50% and <100%
* Syntax score < 32

Exclusion Criteria:

General Exclusion Criteria

* Known hypersensitivity/contraindication to aspirin, heparin or bivalirudin, clopidogrel or ticlopidine, cobalt, nickel, chromium, molybdenum, or sensitivity to contrast media, which can't be adequately pre-medicated
* Platelet count <100,000 cells/mm³ or >700,000 cells/mm³, or a white blood cell (WBC) count <3,000 cells/mm³ within 7 days prior to index procedure
* Serum creatinine level >170 micromol/L within 7 days prior to index procedure
* Evidence of acute MI within 72 hours of intended trial procedure (defined as: QWMI or NQWMI having CK enzymes >2X laboratory upper limit of normal in the presence of a confirming cardiac specific biomarker (Troponin I or T)
* Previous stenting anywhere in target vessel
* Percutaneous coronary intervention (PCI) of non-target vessel within 30 days prior to procedure that results in any MAC(C)E event. If non target vessel stent is implanted within 72 hours prior to index procedure, 2 post procedural serial CK or CK-MB measurements must be below investigational site's upper limit of normal
* PCI of non-target vessel within 24 hours prior to procedure
* Planned PCI of the target vessel within 6 months post-procedure
* During index procedure, target lesion requires treatment with device other than PTCA or cutting balloon prior to stent placement
* Documented left ventricular ejection fraction (LVEF) <30% at most recent evaluation
* History of stroke or transient ischemic attack (TIA) within prior 6 months
* Active peptic ulcer or upper gastrointestinal (GI) bleeding within prior 6 months
* History of bleeding diathesis or coagulopathy or will refuse blood transfusions
* Concurrent medical condition with life expectancy <12 months
* Currently participating in investigational drug or device trial that's not completed the primary endpoint or that clinically interferes with current trial endpoints; or requires coronary angiography, IVUS or other coronary artery imaging procedures.

Angiographic Exclusion Criteria

* Target lesion located in native vessel with saphenous vein graft or left/right internal mammary artery (LIMA/RIMA) bypass
* Target lesion has any of following characteristics:
* Severely calcified
* Evidence of thrombus
* Syntax score ≥33

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2009-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
A composite of cardiac death, target vessel myocardial infarction (MI) and clinically driven target lesion revascularization (TLR) at 30 days post procedure | 30 days (plus or minus 3 days)
  A composite of cardiac death, target vessel myocardial infarction (MI) and clinically driven target lesion revascularization (TLR) at 30 days post procedure.

SECONDARY OUTCOMES:
Angiographic and Procedural success | 30 days (plus or minus 3 days)
  Acute device success, Technical Success, Clinical Procedural Success, Device malfunctions, Ease-of-Use parameters, Main branch and side branch angiographic endpoints, Main branch and side branch IVUS endpoints (Reference Lumen Area; Reference EEM Area; Lesion Lumen Area; Lesion EEM Area; Maximum Atheroma Thickness; Minimum Atheroma Thickness; Lesion Maximum Lumen Diameter; Lesion Minimum Lumen Diameter and derived Measurements; calcium measurement)
Total volume of contrast used | 24 hours
  Total volume of contrast used, in mL
Total index PCI procedure time | 24 hours
  Total index PCI procedure time, in minutes
Target vessel revascularization (TVR) rate | 9 months
  Target vessel revascularization (TVR) rate, at 9 months
Target lesion revascularization (TLR) rate | 9 months
  Target lesion revascularization (TLR) rate, at 9 months
Major Adverse Cardiac and Cerebrovascular Events (MAC(C)E) rate | 9 months
  Major Adverse Cardiac and Cerebrovascular Events (MAC(C)E) rate, at 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Tarantini, MD, Ph.D., Principal Investigator — University of Padua, Department of Cardiac, Thoracic and Vascular Sciences
Locations (6):
- Italy (6):
  - Castelfranco Veneto's Hospital, Castelfranco Veneto
  - Conegliano's Hospital, Conegliano
  - Angel's Hospital, Mestre
  - Mirano's Hospital, Mirano
  - Department of Cardiac, Thoracic and Vascular Sciences, University of Padua, Italy, Padua
  - Vicenza's Hospital, Vicenza

REFERENCES:
- [Derived] Tarantini G, La Vecchia L, Galli M, Favero L, D'Amico G, Buja P, Russo F, Cabianca E, Napodano M, Musumeci G, Franceschini E, Grassi G, Pavei A, Bonmassari R, Cernetti C, Spedicato L, Caprioglio F, Reimers B, Isabella G. Clinical outcome of patients with de novo coronary bifurcation lesions treated with the Tryton Side Branch Stent. The SAFE-TRY prospective multicenter single arm study. Int J Cardiol. 2013 Oct 15;168(6):5323-8. doi: 10.1016/j.ijcard.2013.08.008. Epub 2013 Aug 16. PMID 24007969